CLINICAL TRIAL: NCT00600093
Title: Perioperative Treatment of Parkinsonian Patients With Parenteral Amantadine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI leaving the institute for a fellowship.
Sponsor: Rabin Medical Center (Other)
Responsible Party: Aeyal Raz, MD, PhD, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4332
Record Dates: First submitted 2008-01-13; First posted 2008-01-24 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Parkinson Disease; Perioperative Care
Keywords: Amantadine
MeSH Terms: conditions — Parkinson Disease | interventions — Amantadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Amantadine

INTERVENTIONS:
Drug: Amantadine — IV Amantadine 200mg *1/d at the beginning of surgery and 24 hours following surgery
  Other Names: PK MERZ

SUMMARY:
The purpose of this study is to determine whether administrating of Amantadine (a dopamine agonist) to patients suffering from Parkinson disease during the perioperative period is safe, and to asses potential benefits of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of Parkinson Disease refered for surgery at our institution.

Exclusion Criteria:

* Cardiac and neurosurgical procedures
* Inability to sign informed Consent
* allergy to Amantadine
* Congestive heart failure
* Arrythmia (including bradycardia below 55 bpm)
* renal failure (creatinin above 1.5)
* If a patient will develop agitation or delirium lasting longer then 8 hours he will not receive the second dose of amantadine.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Mortality, Surgical site infection, Pneumonia, Myocardial Infarction, Cerebral Vascular Accident (CVA). | 28 days

SECONDARY OUTCOMES:
UPDRS score | 2,28 days
Pain (vas score), Analgetic drugs requirement | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Aeyal Raz, MD,PhD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Derived] Raz A, Lev N, Orbach-Zinger S, Djaldetti R. Safety of perioperative treatment with intravenous amantadine in patients with Parkinson disease. Clin Neuropharmacol. 2013 Sep-Oct;36(5):166-9. doi: 10.1097/WNF.0b013e31829bd066. PMID 24045608